CLINICAL TRIAL: NCT02436902
Title: Adjuvant Transarterial Chemoembolization With or Without Sorafenib for Patients With Hepatocellular Carcinoma and Microvascular Invasion
Brief Title: Adjuvant Therapies for Patients With HCC and MVI
Acronym: A-TACE/S-HCC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jian-Hong Zhong, Guangxi Medical University, Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-TACE/S-HCC
Record Dates: First submitted 2015-04-28; First posted 2015-05-07 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TACE (Experimental): Transarterial chemoembolization (TACE) is performed two to four weeks after hepatic resection.
  Interventions: Procedure: TACE; Other: empty control
- sorafenib (Active Comparator): Patients will receive sorafenib at a dose of 400 mg twice daily after 2 weeks of hepatic resection.
  Interventions: Drug: Sorafenib
- TACE plus sorafenib (Other): Patients will receive sorafenib at a dose of 400 mg twice daily after 2 weeks of hepatic resection. At the same time, TACE is performed two to four weeks after hepatic resection.
  Interventions: Drug: TACE plus sorafenib; Other: empty control
- empty control (No Intervention): This group patients will receive best supportive care.

INTERVENTIONS:
Procedure: TACE — TACE is performed one month after resection.
  Other Names: transarterial chemoembolization
  Arms: TACE
Drug: Sorafenib — Sorafenib is submitted one month after resection.
  Arms: sorafenib
Drug: TACE plus sorafenib — TACE plus sorafenib will be submitted one month after resection.
  Arms: TACE plus sorafenib
Other: empty control — This group will not receive adjuvant therapy.
  Arms: TACE; TACE plus sorafenib

SUMMARY:
Hepatocellular carcinoma (HCC) is a common malignancy, and its incidence is expected to increase in many countries in coming decades. Though prognosis for patients with HCC is generally poor, hepatic resection can be an effective curative treatment, and its indications have been expanding in recent years. Resection can be reasonably safe and effective even for patients with micro- or macrovascular invasion. However, the recurrence rate of HCC is as high as 74% for patients with intermediate and advanced HCC after resection. Microvascular invasion is one of the main risk factors which influence risk of HCC recurrence and patient prognosis after resection. Therefore, adjuvant therapy to prevent tumor recurrence after resection is so important to improve patient prognosis.

Nowadays, adjuvant transarterial chemoembolization (TACE) is reported to be effective in reducing early recurrence rate and mortality for patients with HCC with risk factors of recurrence. Sorafenib is a novel drug which is effective for advanced stage HCC. However, the efficacy of adjuvant sorafenib for postoperative HCC is unknown. Therefore, it is interesting to investigate the efficacy of adjuvant sorafenib, and compare its efficacy to TACE, TACE plus sorafenib, or best supportive care for patients with postoperative HCC and microvascular invasion.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Diagnosis of HCC was confirmed by histopathological examination of surgical samples in all patients
* Patients with microvascular invasion by histopathological examination of surgical samples
* Patients have Child-Pugh A or B liver function
* No previous neoadjuvant treatment
* No evidence of macrovascular invasion, metastasis to the lymph nodes and/or distant metastases on the basis of preoperative imaging results and perioperative findings
* No malignancy other than HCC for 5 years prior to the initial HCC treatment

Exclusion Criteria:

* History of cardiac disease
* Known history of human immunodeficiency virus (HIV) infection
* Known Central Nervous System tumors including metastatic brain disease
* History of organ allograft
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study
* Pregnant or breast-feeding patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-08-23 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Overall survivals | 1 year

SECONDARY OUTCOMES:
Hospital mortality | 30-day
Recurrence rates | 1 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hepatobilliary Surgery, Affiliated Tumor of Guangxi University, Nanning, Guangxi, China

REFERENCES:
- [Background] Zhong JH, Li LQ. Postoperative adjuvant transarterial chemoembolization for participants with hepatocellular carcinoma: A meta-analysis. Hepatol Res. 2010 Oct;40(10):943-53. doi: 10.1111/j.1872-034X.2010.00710.x. PMID 20887328
- [Background] Llovet JM, Ricci S, Mazzaferro V, Hilgard P, Gane E, Blanc JF, de Oliveira AC, Santoro A, Raoul JL, Forner A, Schwartz M, Porta C, Zeuzem S, Bolondi L, Greten TF, Galle PR, Seitz JF, Borbath I, Haussinger D, Giannaris T, Shan M, Moscovici M, Voliotis D, Bruix J; SHARP Investigators Study Group. Sorafenib in advanced hepatocellular carcinoma. N Engl J Med. 2008 Jul 24;359(4):378-90. doi: 10.1056/NEJMoa0708857. PMID 18650514
- [Background] Zhou L, Rui JA, Wang SB, Chen SG, Qu Q. Early recurrence in large hepatocellular carcinoma after curative hepatic resection: prognostic significance and risk factors. Hepatogastroenterology. 2014 Oct;61(135):2035-41. PMID 25713907